CLINICAL TRIAL: NCT04094792
Title: Depression, Trauma, and Health (DepTH): Efficacy of an mHealth App for Symptom Self-Management in College Students
Brief Title: Depression, Trauma, and Health: Efficacy of an mHealth App for Symptom Self-Management in College Students
Acronym: DepTH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI moving to another university--study will not be done at UK; Coronavirus pandemic will likely delay start at University of Texas at Arlington
Sponsor: Donna Schuman (Other)
Collaborators: Happify Inc. (Industry); University of Kentucky (Other)
Responsible Party: Sponsor-Investigator, Donna Schuman, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 53054
Record Dates: First submitted 2019-09-16; First posted 2019-09-19 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Depression
Keywords: heart rate variability; autonomic function; biofeedback; mobile health
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: two-group randomized controlled efficacy trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intervention (Experimental): For the intervention group, baseline measures on depression and heart rate variability will be obtained at baseline and post-test (21 days later). Intervention group subjects will use the Breather app twice daily, five minutes each time, for a period of 21 days.
  Interventions: Device: Happify Breather App
- Control (No Intervention): For the control group, baseline measures on depression and heart rate variability will be obtained at baseline and post-test (21 days later).

INTERVENTIONS:
Device: Happify Breather App — Subjects in the intervention group will be cued to breathe at 6 breaths per minute and will receive real time heart rate variability biofeedback. As they increase HRV, screen elements will become more visually appealing.
  Arms: Intervention

SUMMARY:
The study is designed to examine the efficacy of a mobile application heart rate variability biofeedback exercise on heart rate variability and depression.

The main objective of this study is to assess the Breather app manufactured by Happify, Inc., as a tool for improving levels of depression and heart rate variability in college students.Happify™ Breather is a mobile app that provides users with HRV biofeedback aimed at improving mental health and wellness. Breather uses HRV sensors to help users control breathing, leading to calm and relaxation. The more relaxed users are, the more visually reinforcing scene elements will appear in the underwater environment of the game. Breather uses an optical sensor in a smartphone camera. During app use, users are cued by the app to breathe at 6 cycles/minute using a breath pacer. When the smartphone camera flash is illuminated, color signal changes are measured from the fingertip pressed to the camera lens.

The study population is college students who score in the clinical range on the PHQ-9. Secondary outcomes include anxiety, somatoform symptoms, and app adherence.

DETAILED DESCRIPTION:
Although traditionally considered a healthy group, concern is mounting about the health and mental health of college students (Hunt & Eisenberg, 2010). Mental health problems, such as depression, often go untreated in young college-age adults (Saeb et al., 2015). Depression is associated with poor health outcomes (Rutter et al., 2013). Suicide, often associated with depression, is a leading cause of death in college students (Drapeau & McIntosh, 2015). Research suggests that stress-related interventions would be useful for college students at risk of poor mental health outcomes (Karatekin, 2017); however less is known about the impact of mobile health interventions on depression in college students.

Studies have shown that heart rate variability (HRV), a potent all-cause morbidity and mortality indicator, is reduced in persons with depressive disorders (Kemp, Quintana, Felmingham, Matthews, & Jelinek, 2012). Although HRV is typically higher in college-age students because they are often younger, studies have shown that college students HRV biofeedback involves voluntary changes in breathing rate, rhythm, pattern, and quality. Within a few minutes of rhythmic stimulation of the cardiovascular system through slow paced breathing at around six breaths per minute, HRV biofeedback produces robust increases in HRV (Vaschillo, Vaschillo, & Lehrer, 2006). Emotional regulation, to include depressive symptoms, can be improved through HRV biofeedback (Henriques, Keffer, Abrahamson, & Horst, 2011; Siepmann, Aykac, Unterdörfer, Petrowski, & Mueck-Weymann, 2008).

Smart phones offer an expedient way to deliver digital interventions that promote relaxation and improve mood. Happify™ Breather is a mobile app that provides users with HRV biofeedback aimed at improving mental health and wellness. Breather uses HRV sensors to help users control breathing, leading to calm and relaxation. The more relaxed users are, the more visually reinforcing scene elements will appear in the underwater environment of the game. Breather uses an optical sensor in a smartphone camera. During app use, users are cued by the app to breathe at 6 cycles/min using a breath pacer. When the smartphone camera flash is illuminated, red color signal changes (increasing with systole and decreasing with diastole) are measured from the fingertip pressed to the camera lens and sampled at 50 Hz. In a validation study, results obtained from the Happify™ HRV biofeedback Breather app were consistent with Holter monitor results (Stein, 2018). The app is free of charge and publicly available on the iTunes App Store.

The primary objective of the study is to examine the efficacy of the Happify™ Breather app's biofeedback exercise in improving high frequency (HF) heart rate variability (HRV) measures and depression scores in students compared to control. Secondary outcomes are to test the efficacy of the app for anxiety and somatoform symptoms, as well as adherence to the app.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45;
* University of Kentucky college student;
* Self-reported low mood;
* Own a smart phone or iPod (6th Generation or later).

Exclusion Criteria:

* Score >/= 10 on the PHQ-9 measure from the PHQ-SADS;
* Self-reported diagnosis of lung disease (e.g., Chronic Obstructive Pulmonary - Disease. Asthma requiring medication), coronary heart disease, stroke, or uncontrolled diabetes (HA1c>7.0);
* Self-reported history or diagnosis of seizure disorder;
* Self-reported prescription for tricyclic antidepressants and/or clozapine
* Current smoking or vaping (use in last 30 days);
* Previous participation in an HRV biofeedback study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-05 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Depression | 3 weeks
  Change in scores on the Patient Health Questionnaire-9 (PHQ-9) from baseline to week 3
Low Frequency HRV | 3 weeks
  Change from baseline to week 3 measured by electrocardiogram
High Frequency HRV | 3 weeks
  Change from baseline to week 3 measured by electrocardiogram

SECONDARY OUTCOMES:
Anxiety | 3 weeks
  Change from baseline to week 3 measured by scores on the GAD-7 (Generalized Anxiety Disorder-7)
Heart Rate Variability Low Frequency/High Frequency Ratio | 3 weeks
  Change from baseline to week 3 measured by electrocardiogram
Somatoform | 3 weeks
  Change from baseline to week 3 measured by scores on the PHQ-15 (Patient Health Questionnaire-15)
App Adherence | 3 weeks
  Number of times app is used over 21 days

CONTACTS AND LOCATIONS:
Locations (1):
- Donna L. Schuman, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No